CLINICAL TRIAL: NCT05187403
Title: A Placebo-Controlled, Double-masked Phase-1 Study in Healthy Subjects Investigating the Safety and Tolerability of Laquinimod Eye Drops
Brief Title: A Study of Laquinimod Eye-drops in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 21LAQ01; 2021-004029-60 (EudraCT Number)
Record Dates: First submitted 2021-12-06; First posted 2022-01-11 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Laquinimod - Single Ascending Doses (Experimental): One single dose of laquinimod eye-drops. There are up to four planned dose levels.
  Interventions: Drug: Laquinimod
- Placebo - Single Ascending Doses (Placebo Comparator): One single dose of placebo eye-drops.
  Interventions: Drug: Placebo
- Laquinimod - Multiple Ascending Doses (Experimental): Eye-drops administered once daily for 14-21 days. There are up to two planned dose levels. The first dose level will be defined in the SAD-part of the study.
  Interventions: Drug: Laquinimod
- Placebo - Multiple Ascending Doses (Placebo Comparator): Eye-drops administered once daily for 14-21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Laquinimod — Eye-drops
  Other Names: TV-5600; ABR-215062
  Arms: Laquinimod - Multiple Ascending Doses; Laquinimod - Single Ascending Doses
Drug: Placebo — Eye-drops
  Arms: Placebo - Multiple Ascending Doses; Placebo - Single Ascending Doses

SUMMARY:
This is a Phase 1 randomized, double-masked, placebo-controlled study performed with healthy participants to assess the safety and tolerability of laquinimod eye-drops.

DETAILED DESCRIPTION:
Laquinimod administered as an oral capsule formulation has previously been studied in neurodegenerative and autoimmune diseases. The clinical side effect profile of orally administered laquinimod is well-characterized based on this previous experience.

This trial will establish a safe and tolerated dose of laquinimod when administered as an eye-drop formulation following single ascending dose (SAD) and multiple ascending dose (MAD) administrations. There are four planned groups in the SAD-part of the study which will enroll 28 participants, if all dose levels are explored. The subsequent MAD-part of the study will enroll another 28 participants.

ELIGIBILITY:
Main inclusion criteria:

* In good health according to medical history, physical examination, vital signs, ECG and clinical chemistry, urinary and hematological laboratory tests

Main exclusion criteria:

* Unable or unwilling to use eye-drops
* Current usage of contact lenses
* History of eye surgery
* Sign or symptom of active eye disease
* History of an eye disease or other condition that could interfere with eye examinations in the study, or with ocular absorption of the investigational product
* History of inflammatory ocular disease
* History of cardiovascular or pulmonary disorder
* Family history of known or suspected hereditary cardiovascular disease
* Autoimmune disease or known family history of autoimmune disease
* Any other condition that would contraindicate subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Adverse events | For 7 days post-dose
  Type, frequency, seriousness, severity and relationship to treatment

SECONDARY OUTCOMES:
Participant-reported eye-toxicities | Pre-dose (baseline) and immediately after the intervention
  Assessed from change from baseline in ocular symptoms score determined using a Visual Analogue Scale with 0-100 range, where 0= no symptom and 100= worst possible discomfort.
Investigator-reported eye-toxicities - BCVA | Pre-dose (baseline) and immediately after the intervention
  Assessed from change from baseline in Best Corrected Visual Acuity (BCVA) using the Early Treatment Diabetic Retinopathy Study research group (ETDRS) visual acuity chart with objective and subjective refraction.
Investigator-reported eye-toxicities - Slit lamp examination | Pre-dose (baseline) and immediately after the intervention
  Assessed from change from baseline in slit lamp examination parameters (eyelid swelling, eyelid redness, conjunctival redness, conjunctival chemosis, scleral redness, corneal opacity, iris alterations and anterior chamber flare) graded on a 4-point scale where 0= none, 1= mild, 2= moderate, and 3= severe.
Investigator-reported eye-toxicities - Corneal fluorescein staining | At screening visit (baseline) and immediately after the intervention
  Assessed from change from baseline in corneal fluorescein staining determined using the NEI/Industry Workshop guidelines. The cornea is divided into five sectors (central, superior, inferior, nasal and temporal) and each sector scored on a 4-point scale, where 0= no staining and 3= maximum staining.
Investigator-reported eye-toxicities - Intraocular pressure | At screening visit (baseline) and immediately after the intervention
  Assessed from change from baseline in intraocular pressure (mmHg) determined using a Goldmann applanation tonometer.
Investigator-reported eye-toxicities - Funduscopy in mydriasis | At screening visit (baseline) and immediately after the intervention
  Assessed from change from baseline in clinical signs detected by indirect funduscopic inspection of the optic disc, macula, retinal vessels and retinal periphery.
Peak plasma concentration of laquinimod | Over up to 21 days after (last) dose
  Maximal plasma concentration (Cmax) of laquinimod as assessed from samples collected pre-dose and at frequent intervals over 7 days after (last) dose
Time to peak plasma concentration of laquinimod | Over up to 21 days) after (last) dose
  Time to maximal plasma concentration (tmax) of laquinimod as assessed from samples collected pre-dose and at frequent intervals over 7 days after (last) dose
Trough plasma concentration of laquinimod at steady-state | On the last three days of multiple dosing
  Minimal plasma concentration (Cmin,ss) of laquinimod as assessed from samples collected pre-dose on Days 12, 13 and 14 within the multiple-dose arm
Systemic exposure of laquinimod | Over up to 21 days after (last) dose
  Area under the plasma concentration time curve (AUC) of laquinimod

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD PhD, Principal Investigator — Clinical trial center at Medical University Vienna
Locations (1):
- Clinical trial center at Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No